CLINICAL TRIAL: NCT05616013
Title: A Randomized, Double-Blind, Placebo-Controlled Multi-Center Study of Intravenous Bimagrumab, Alone or in Addition to Open Label Subcutaneous Semaglutide, to Investigate the Efficacy and Safety in Overweight or Obese Men and Women
Brief Title: Safety and Efficacy of Bimagrumab and Semaglutide in Adults Who Are Overweight or Obese
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Versanis Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 18828; J4Z-MC-GIDA (Other: Eli Lilly and Company); VER201-PH2-031 (Other: Versanis)
Record Dates: First submitted 2022-10-16; First posted 2022-11-14 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Obese; Overweight or Obesity
Keywords: bimagrumab; semaglutide
MeSH Terms: conditions — Obesity; Overweight | interventions — bimagrumab; semaglutide

STUDY DESIGN:
Intervention Model Description: The study is designed to have three periods. The 48-week core treatment period has 9 treatment arms, with combinations of 3 semaglutide doses (none, 1.0 mg and 2.4 mg) and 3 bimagrumab doses (0, 10 and 30 mg/kg). The core treatment period is then followed by an open-label 24-week treatment extension period during which participants originally assigned to either placebo or bimagrumab 10 mg/kg will switch to bimagrumab 30 mg/kg. All other treatment assignments will remain the same. The extension period is then followed by a 32-week post-treatment period, during which all study treatments will be withdrawn from all arms.
Who Masked: Participant, Investigator
Masking Description: In regard to bimagrumab and placebo-bimagrumab, the participants, Investigator and Sponsor will be blinded.
  Due to semaglutide being pre-filled, packaged and labeled by manufacturer, it is not possible to blind semaglutide.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Placebo (Placebo Comparator): Participants received a placebo administered intravenously (IV) at baseline and at weeks 4, 16, 28, and 40 during the core treatment period.
  Interventions: Other: Placebo
- Bimagrumab 10 mg/kg (Experimental): Participants received bimagrumab 10 milligrams/kilogram (mg/kg) administered IV at baseline and at weeks 4, 16, 28, and 40 during the core treatment period.
  Interventions: Biological: Bimagrumab
- Bimagrumab 30 mg/kg (Experimental): Participants received bimagrumab 30 mg/kg administered IV at baseline and at weeks 4, 16, 28, and 40.
  Interventions: Biological: Bimagrumab
- Placebo + Semaglutide 1.0 mg (Experimental): Participants received a placebo administered IV at baseline and at Weeks 4, 16, 28, and 40, and 1 milligram (mg) of semaglutide administered subcutaneously (SC) weekly for 48 weeks as per the below dose escalation schedule:
  Weeks 1 to 4: 0.25 mg Weeks 5 to 8: 0.5 mg Weeks 9 to 48: 1.0 mg
  Interventions: Drug: Semaglutide; Other: Placebo
- Placebo + Semaglutide 2.4 mg (Experimental): Participants received a placebo administered IV at baseline and at weeks 4, 16, 28, and 40, and 2.4 mg semaglutide administered SC weekly for 48 weeks as per the below dose escalation schedule:
  Weeks 1 to 4: 0.25 mg Weeks 5 to 8: 0.5 mg Weeks 9 to 12: 1.0 mg Weeks 13 to 16: 1.7 mg Weeks 17 to 48: 2.4 mg.
  Interventions: Drug: Semaglutide; Other: Placebo
- Bimagrumab 10 mg/kg + Semaglutide 1.0 mg (Experimental): Participants received bimagrumab 10 mg/kg administered IV at baseline and at weeks 4, 16, 28, and 40, and 1 mg semaglutide administered SC weekly for 48 weeks as per the below dose escalation schedule:
  Weeks 1 to 4: 0.25 mg Weeks 5 to 8: 0.5 mg Weeks 9 to 48: 1.0 mg.
  Interventions: Biological: Bimagrumab; Drug: Semaglutide
- Bimagrumab 10 mg/kg + Semaglutide 2.4 mg (Experimental): Participants received bimagrumab 10 mg/kg administered IV at baseline and at weeks 4, 16, 28, and 40, and 2.4 mg semaglutide administered SC weekly for 48 weeks as per the below dose escalation schedule:
  Weeks 1 to 4: 0.25 mg Weeks 5 to 8: 0.5 mg Weeks 9 to 12: 1.0 mg Weeks 13 to 16: 1.7 mg Weeks 17 to 48: 2.4 mg.
  Interventions: Biological: Bimagrumab; Drug: Semaglutide
- Bimagrumab 30 mg/kg + Semaglutide 1.0 mg (Experimental): Participants received bimagrumab 30 mg/kg administered IV at baseline and at weeks 4, 16, 28, and 40, and 1 mg semaglutide administered SC weekly for 48 weeks as per the below dose escalation schedule:
  Weeks 1 to 4: 0.25 mg Weeks 5 to 8: 0.5 mg Weeks 9 to 48: 1.0 mg
  Interventions: Biological: Bimagrumab; Drug: Semaglutide
- Bimagrumab 30 mg/kg + semaglutide 2.4 mg (Experimental): Participants received bimagrumab 30 mg/kg administered IV at baseline and at weeks 4, 16, 28 and 40, and 2.4 mg semaglutide administered SC weekly for 48 weeks as per the below dose escalation schedule:
  Weeks 1 to 4: 0.25 mg Weeks 5 to 8: 0.5 mg Weeks 9 to 12: 1.0 mg Weeks 13 to 16: 1.7 mg Weeks 17 to 48: 2.4 mg.
  Interventions: Biological: Bimagrumab; Drug: Semaglutide

INTERVENTIONS:
Biological: Bimagrumab — Human monoclonal antibody to the activin receptor type II
  Arms: Bimagrumab 10 mg/kg; Bimagrumab 10 mg/kg + Semaglutide 1.0 mg; Bimagrumab 10 mg/kg + Semaglutide 2.4 mg; Bimagrumab 30 mg/kg; Bimagrumab 30 mg/kg + Semaglutide 1.0 mg; Bimagrumab 30 mg/kg + semaglutide 2.4 mg
Drug: Semaglutide — Glucagon-like peptide-1 (GLP-1) receptor agonist
  Other Names: Wegovy; Ozempic
  Arms: Bimagrumab 10 mg/kg + Semaglutide 1.0 mg; Bimagrumab 10 mg/kg + Semaglutide 2.4 mg; Bimagrumab 30 mg/kg + Semaglutide 1.0 mg; Bimagrumab 30 mg/kg + semaglutide 2.4 mg; Placebo + Semaglutide 1.0 mg; Placebo + Semaglutide 2.4 mg
Other: Placebo — Placebo
  Arms: Placebo; Placebo + Semaglutide 1.0 mg; Placebo + Semaglutide 2.4 mg

SUMMARY:
A phase 2 study to assess the efficacy of bimagrumab alone or in addition to semaglutide to assess efficacy and safety in overweight or obese men and women

DETAILED DESCRIPTION:
This study investigates if bimagrumab in addition to semaglutide is able to preserve/increase muscle mass in the presence of weight and/or fat mass loss.

ELIGIBILITY:
Key Inclusion Criteria:

* A written informed consent must be obtained before any study-related assessments are performed.
* Men and women between 18 and 80 years, inclusive; women of child-bearing potential (defined as those who are not post-menopausal or post-surgical sterilization) must meet both of the following criteria:

  * Two negative pregnancy tests (at screening and at randomization, prior to dosing)
  * Use of intrauterine device, from at least 3 months before the baseline visit through at least 4 months after the last dose of bimagrumab/placebo i.v., and an additional contraceptive (barrier) method from screening through at least 4 months after the last dose of bimagrumab/placebo i.v.
* Body mass index (BMI) ≥ 30 or BMI ≥ 27 with one or more obesity-associated comorbidities (e.g., hypertension, insulin resistance, sleep apnea, or dyslipidemia)
* Stable body weight (± 5 kg) within 90 days of screening, and body weight <150 kg
* Have a history of at least one self-reported unsuccessful behavioral effort to lose body weight
* Able to communicate well with the Investigator, comply with the study requirements and adhere to the diet and activity programs for the study duration

Key Exclusion Criteria:

* History of, or known hypersensitivity to, monoclonal antibody drugs or a contraindication to semaglutide (Ozempic® or Wegovy®)
* Use of other investigational drugs at the time of enrollment or within 30 days or 5 half-lives of enrollment, whichever is longer, or longer if required by local regulations
* Treatment with any medication for the indication of obesity within the past 30 days before screening
* Diagnosis of diabetes requiring current use of any antidiabetic drug or HbA1c ≥ 6.5% Note: Metabolic syndrome is not an exclusion, even if managed with an anti-diabetic drug such as metformin or an SGLT2 inhibitor. A diagnosis of prediabetes or impaired glucose tolerance managed exclusively with non-pharmacologic approaches (e.g., diet and exercise) is not an exclusion.
* Any chronic infections likely to interfere with study conduct or interpretation such as hepatitis B (HBV), hepatitis C (HCV), or human immunodeficiency virus (HIV). History of hepatitis A or hepatitis C successfully treated is not exclusionary. Active COVID-19 infection.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to initial dosing, or longer if required by local regulation, or plasma donation (> 250 mL) within 14 days prior to the first dose
* Any disorder, unwillingness, or inability not covered by any of the other exclusion criteria, which in the Investigator's opinion, might jeopardize the participant's safety or compliance with the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2025-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (26):
- United States (10):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - Altus Research, Lake Worth, Florida
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Weill Cornell Medical College, New York, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - SPICA Clinical, Columbia, South Carolina
  - Mt. Olympus Medical Research, Sugar Land, Texas
- Australia (8):
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - University of The Sunshine Coast Morayfield, Morayfield, Queensland
  - University of the Sunshine Coast Clinical Trial Centre, Sippy Downs, Queensland
  - University of The Sunshine Coast South Brisbane, South Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Austin Health, Heidelberg Heights, Victoria
  - Emeritus Research, Camberwell
- New Zealand (8):
  - Southern Clinical Trials Ltd, Beckenham, Christchurch, Canterbury
  - P3 Research, Newtown, Wellington Region
  - New Zealand Clinical Research Auckland, Auckland
  - Optimal Clinical Trials, Auckland
  - Middlemore Hospital, Auckland
  - New Zealand Clinical Research Christchurch, Christchurch
  - Lakeland Clinical Trials Waikato, Hamilton
  - Southern Clinical Trials Tasman, Nelson

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Moon S, Choi JW, Park JH, Kim DS, Ahn Y, Kim Y, Kong SH, Oh CM. Association of Appendicular Skeletal Muscle Mass Index and Insulin Resistance With Mortality in Multi-Nationwide Cohorts. J Cachexia Sarcopenia Muscle. 2025 Apr;16(2):e13811. doi: 10.1002/jcsm.13811. PMID 40230053

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was designed to be conducted in three phases: Core Treatment period (Weeks 1 to 48) followed by Open Label Extension Treatment Period (Weeks 49 to 72) and Post-Treatment Follow-Up Period (Weeks 73 to 104) Currently, only the results from the Core Treatment phase (up to Week 48) are available. Data from Open Label Extension (up to Week 72) and Post-Treatment Follow-Up (up to Week 104) are still being analyzed and will be reported at the time of final results reporting by June 2026.
Groups:
- Placebo + Semaglutide 1.0 mg: Participants received a placebo administered IV at baseline and at Weeks 4, 16, 28, and 40, and 1 milligram (mg) of semaglutide administered subcutaneously (SC) weekly for 48 weeks as per the below dose escalation schedule:
  Weeks 1 to 4: 0.25 mg Weeks 5 to 8: 0.5 mg Weeks 9 to 48: 1.0 mg
  .
Period: Overall Study
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Started | 56 | 56 | 57 | 56 | 57 | 56 | 56 | 56 | 57
Safety Analysis Population (Received at Least 1 Dose of Study Drug) | 55 | 56 | 57 | 55 | 56 | 56 | 55 | 56 | 55
Completed ("Completed" includes participants who completed the study until Week 48 and were moved to the other treatment periods. Open Label Extension Treatment Period (Weeks 49 to 72) and Post-Treatment Follow-Up Period (Weeks 73 to 104) analyses are ongoing and will be presented at the time of reporting the final results.) | 29 | 27 | 33 | 40 | 48 | 36 | 39 | 43 | 42
Not Completed | 27 | 29 | 24 | 16 | 9 | 20 | 17 | 13 | 15
Not completed — Adverse Event | 6 | 12 | 8 | 4 | 6 | 8 | 3 | 6 | 1
Not completed — Lost to Follow-up | 5 | 4 | 3 | 2 | 0 | 5 | 2 | 1 | 2
Not completed — Non-compliance with study requirements | 2 | 2 | 2 | 3 | 0 | 2 | 1 | 1 | 4
Not completed — Withdrawal by Subject | 11 | 9 | 8 | 6 | 3 | 4 | 6 | 5 | 4
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Did not Fulfill Enrollment criteria | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Difficulty Attending Visits due to Personal/work Commitments | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Withdrawal due to use of Restricted Medication | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Cannot Continue study due to Work Commitments | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Decision, Time Constraints | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Prohibited Concomitant Medication | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Medical history condition Requiring Further Treatment | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Difficulty Following Protocol Requirement, Dissatisfied with Amount of Weight Lost | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawn due to Elevated Blood Pressure | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant Reported Concerns About their fat Percentage Dropping too low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Unable to Visit site as Participant Moved town | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg | Total
Number analyzed (Participants) | 56 | 56 | 57 | 56 | 57 | 56 | 56 | 56 | 57 | 507
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (14.6) | 44.4 (10.9) | 49.2 (12.2) | 50.3 (11.2) | 49.6 (11.8) | 44.8 (12.0) | 46.2 (11.7) | 47.7 (10.4) | 47.5 (12.7) | 47.5 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 33 | 32 | 33 | 32 | 32 | 32 | 33 | 291
  Male | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 216
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 11 | 3 | 4 | 2 | 5 | 7 | 7 | 8 | 53
  Not Hispanic or Latino | 48 | 44 | 53 | 52 | 54 | 50 | 49 | 47 | 48 | 445
  Unknown or Not Reported | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  Asian | 1 | 1 | 1 | 0 | 3 | 1 | 4 | 1 | 3 | 15
  Black | 6 | 3 | 4 | 7 | 5 | 7 | 5 | 6 | 3 | 46
  Native Hawaiian or Other Pacific Islander | 5 | 3 | 2 | 1 | 1 | 2 | 6 | 3 | 1 | 24
  Other | 4 | 2 | 4 | 3 | 1 | 1 | 2 | 3 | 3 | 23
  White | 38 | 44 | 45 | 40 | 46 | 41 | 39 | 43 | 45 | 381
  Multiple | 2 | 2 | 0 | 4 | 1 | 4 | 0 | 0 | 0 | 13
  Unknown | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 12 | 8 | 17 | 9 | 19 | 5 | 7 | 14 | 14 | 105
  New Zealand | 24 | 24 | 23 | 26 | 23 | 25 | 30 | 24 | 23 | 222
  United States | 20 | 24 | 17 | 21 | 15 | 26 | 19 | 18 | 20 | 180
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 109.55 (19.33) | 105.12 (19.50) | 109.05 (17.56) | 105.81 (20.02) | 104.50 (14.82) | 108.36 (18.92) | 108.78 (18.41) | 108.19 (14.34) | 108.12 (18.48) | 107.50 (17.97)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Body Weight at Week 48
Description: Least square (LS) Mean was determined by analysis of covariance (ANCOVA) model using Baseline + Gender (Male, Female) + Country (Australia, New Zealand, United States of America) + Treatment (Type III sum of squares) as variables. Only participants with non-missing baseline value were included in analysis. Missing values at Week 48 were imputed 100 times based on observed data in the Placebo arm
Time Frame: Baseline, Week 48
Population: All randomized participants who received at least one dose of the study drug, had a baseline and at least one post- baseline value for this outcome.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 35 | 31 | 37 | 45 | 51 | 41 | 40 | 43 | 43
kilogram (kg) | -3.31 (1.39) | -5.99 (1.42) | -9.25 (1.33) | -9.76 (1.25) | -14.24 (1.17) | -12.73 (1.29) | -14.31 (1.34) | -13.86 (1.29) | -17.79 (1.29)
Statistical Analysis 1: Comparison: Placebo vs Bimagrumab 30 mg/kg + Semaglutide 2.4 mg; Bima 30mg/kg + Sema 2.4mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Change difference = -14.5, 95% CI 2-sided [-18.0 to -11.0]
Statistical Analysis 2: Comparison: Placebo vs Bimagrumab 30 mg/kg + Semaglutide 1.0 mg; Bima 30mg/kg + Sema 1.0mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Change difference = -10.5, 95% CI 2-sided [-14.0 to -7.09]
Statistical Analysis 3: Comparison: Placebo vs Bimagrumab 10 mg/kg + Semaglutide 2.4 mg; Bima 10mg/kg + Sema 2.4mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Change difference = -11.0, 95% CI 2-sided [-14.4 to -7.55]
Statistical Analysis 4: Comparison: Placebo vs Bimagrumab 10 mg/kg + Semaglutide 1.0 mg; Bima 10mg/kg + Sema 1.0mg vs Placebo; Test type: Superiority; p < .001, ANCOVA; LS Mean Change difference = -9.41, 95% CI 2-sided [-12.9 to -5.93]
Statistical Analysis 5: Comparison: Placebo vs Placebo + Semaglutide 2.4 mg; Sema 2.4mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Change difference = -10.9, 95% CI 2-sided [-14.4 to -7.46]
Statistical Analysis 6: Comparison: Placebo vs Placebo + Semaglutide 1.0 mg; Sema 1.0mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Change difference = -6.45, 95% CI 2-sided [-9.96 to -2.94]
Statistical Analysis 7: Comparison: Placebo vs Bimagrumab 30 mg/kg; Bima 30mg/kg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Change difference = -5.94, 95% CI 2-sided [-9.47 to -2.41]
Statistical Analysis 8: Comparison: Placebo vs Bimagrumab 10 mg/kg; Bima 10mg/kg vs Placebo; Test type: Superiority; p = 0.133, ANCOVA; LS Mean Change difference = -2.68, 95% CI 2-sided [-6.18 to 0.82]

2. Secondary Outcome: Change From Baseline in Waist Circumference at Week 48
Description: Waist circumference was measured in standing position with a non-stretchable measuring tape to the nearest 0.1 centimeter (cm). LS Mean was determined by ANCOVA model using Baseline + Gender (Male, Female) + Country (Australia, New Zealand, United States of America) + Treatment (Type III sum of squares) as variables. Only participants with non-missing baseline value were included in analysis. Missing values at Week 48 were imputed 100 times based on observed data in the Placebo arm.
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: centimeter (cm)
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 35 | 31 | 37 | 45 | 51 | 41 | 39 | 43 | 43
centimeter (cm) | -4.62 (1.59) | -7.31 (1.74) | -9.10 (1.49) | -8.74 (1.38) | -12.14 (1.27) | -12.41 (1.48) | -13.35 (1.47) | -13.64 (1.42) | -15.78 (1.40)

3. Secondary Outcome: Change From Baseline in Waist Circumference at Week 72
Description: Waist circumference was measured in standing position with a non-stretchable measuring tape to the nearest 0.1 cm.
Time Frame: Baseline, Week 72
Reporting Status: Not Posted, anticipated posting 2026-06

4. Secondary Outcome: Change From Baseline in Total Body Fat Mass in Kilograms (kg) at Week 48
Description: Fat mass was obtained by Dual energy X-ray absorptiometry (DXA) was used to assess changes in body composition. LS Mean was determined by ANCOVA model using Baseline + Gender (Male, Female) + Country (Australia, New Zealand, United States of America) + Treatment (Type III sum of squares) as variables. Only participants with non-missing baseline value were included in analysis. Missing values at Week 48 were imputed 100 times based on observed data in the Placebo arm.
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 30 | 30 | 36 | 45 | 47 | 42 | 40 | 42 | 43
kg | -1.9 (1.18) | -5.7 (1.19) | -8.6 (1.15) | -6.7 (1.04) | -9.6 (1.02) | -11.2 (1.11) | -11.9 (1.11) | -12.2 (1.08) | -15.6 (1.04)

5. Secondary Outcome: Change From Baseline in Total Body Fat Mass in kg at Week 72
Description: Fat mass was obtained by DXA and was used to assess changes in body composition.
Time Frame: Baseline, Week 72
Reporting Status: Not Posted, anticipated posting 2026-06

6. Secondary Outcome: Change From Baseline in Body Fat Percentage at Week 48
Description: Body fat percentage was obtained by DXA was used to assess changes in body composition. LS Mean was determined by ANCOVA model using Baseline + Gender (Male, Female) + Country (Australia, New Zealand, United States of America) + Treatment (Type III sum of squares) as variables. Only participants with non-missing baseline value were included in analysis. Missing values at Week 48 were imputed 100 times based on observed data in the Placebo arm.
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of body fat
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 30 | 30 | 36 | 45 | 47 | 42 | 40 | 42 | 43
percentage of body fat | -1.02 (0.74) | -3.42 (0.76) | -5.23 (0.70) | -3.27 (0.68) | -4.18 (0.66) | -6.25 (0.69) | -7.13 (0.70) | -7.46 (0.68) | -9.30 (0.67)

7. Secondary Outcome: Change From Baseline in Body Fat Percentage at Week 72
Description: Percent body fat obtained by DXA was used to assess changes in body composition.
Time Frame: Baseline, Week 72
Reporting Status: Not Posted, anticipated posting 2026-06

8. Secondary Outcome: Change From Baseline in Visceral Adipose Tissue (VAT), Subcutaneous Adipose Tissue (SAT) and Trunk Fat Mass by DXA at Week 48
Description: DXA was used to assess changes in body composition. LS Mean was determined by ANCOVA model using Baseline + Gender (Male, Female) + Country (Australia, New Zealand, United States of America) + Treatment (Type III sum of squares) as variables. Only participants with non-missing baseline value were included in analysis. Missing values at Week 48 were imputed 100 times based on observed data in the Placebo arm
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 30 | 30 | 36 | 45 | 47 | 42 | 40 | 42 | 43
kg
  VAT: number analyzed (Participants) | 28 | 30 | 32 | 44 | 45 | 41 | 40 | 41 | 41
  VAT | -0.0 (0.08) | -0.3 (0.08) | -0.4 (0.08) | -0.3 (0.06) | -0.4 (0.07) | -0.5 (0.07) | -0.6 (0.07) | -0.6 (0.07) | -0.7 (0.07)
  SAT: number analyzed (Participants) | 29 | 30 | 34 | 44 | 46 | 41 | 40 | 41 | 41
  SAT | -0.05 (0.10) | -0.37 (0.10) | -0.54 (0.10) | -0.43 (0.09) | -0.64 (0.09) | -0.70 (0.09) | -0.84 (0.09) | -0.81 (0.09) | -1.05 (0.09)
  Trunk fat mass | -0.94 (0.72) | -3.54 (0.72) | -5.44 (0.71) | -3.83 (0.64) | -5.48 (0.63) | -6.69 (0.65) | -7.46 (0.66) | -7.51 (0.65) | -9.19 (0.65)

9. Secondary Outcome: Change From Baseline in VAT, SAT and Trunk Fat Mass by DXA at Week 72
Description: DXA was used to assess changes in body composition.
Time Frame: Baseline, Week 72
Reporting Status: Not Posted, anticipated posting 2026-06

10. Secondary Outcome: Percentage of Participants With Reduction in Waist Circumference ≥ 5 cm at Week 48
Description: Waist circumference was measured in a standing position with a non-stretchable measuring tape to the nearest 0.1 cm.
Time Frame: Week 48
Population: All randomized participants who received at least one dose of the study drug and had evaluable data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 55 | 56 | 57 | 55 | 56 | 56 | 55 | 56 | 55
percentage of participants | 47.1 | 60.5 | 67.6 | 62.6 | 79.3 | 81.9 | 84.5 | 81.6 | 86.5

11. Secondary Outcome: Percentage of Participants With Reduction in Body Weight ≥ 5%, ≥ 10% and ≥15% at Week 48
Description: Body weight was measured in kgs to the nearest 0.1 kg.
Time Frame: Week 48
Population: All randomized participants who received at least one dose of the study drug and had evaluable data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 55 | 56 | 57 | 55 | 56 | 56 | 55 | 56 | 55
percentage of participants
  Reduction in ≥ 5% Body Weight | 38.8 | 51.8 | 68.8 | 67.8 | 88.2 | 82.9 | 84.2 | 83.9 | 86.1
  Reduction in ≥ 10% Body Weight | 10.4 | 25.0 | 39.3 | 43.4 | 74.8 | 54.9 | 72.1 | 66.2 | 79.2
  Reduction in ≥ 15% Body Weight | 5.3 | 11.7 | 23.3 | 30.3 | 43.4 | 32.2 | 41.6 | 47.7 | 63.9

12. Secondary Outcome: Percentage of Participants With Reduction in Fat Mass ≥ 5% ≥ 10% ≥ 15% by DXA at Week 48
Description: DXA was used to assess the changes in body composition.
Time Frame: Week 48
Population: All randomized participants who received at least one dose of the study drug and had evaluable data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 52 | 55 | 55 | 55 | 56 | 56 | 55 | 55 | 54
percentage of participants
  ≥ 5% reduction in Fat Mass | 45.3 | 74.4 | 79.3 | 75.7 | 90.6 | 88.5 | 86.4 | 87.9 | 90.0
  ≥ 10% reduction in Fat Mass | 25.9 | 65.1 | 68.3 | 59.5 | 83.2 | 82.7 | 79.5 | 82.1 | 87.1
  ≥ 15% reduction in Fat Mass | 12.7 | 39.4 | 54.8 | 47.8 | 76.1 | 75.7 | 75.9 | 73.5 | 84.1

13. Secondary Outcome: Percentage of Participants With Reduction in Fat Mass ≥ 10% With <5% Decrease (or an Increase) in Lean Mass by DXA at Week 48
Description: DXA was used to assess changes in body composition.
Time Frame: Week 48
Population: All randomized participants who received at least one dose of the study drug and had evaluable data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 52 | 55 | 55 | 55 | 56 | 56 | 55 | 55 | 54
percentage of participants | 18.1 | 55.9 | 58.3 | 26.3 | 20.4 | 52.6 | 52.9 | 63.7 | 58.9

14. Secondary Outcome: Percentage of Participants Achieving >5 kg Weight Loss and Fat Loss Index (FLI) of >70%, >80%, and >90% by DXA at Week 48
Description: DXA was used to assess changes in body composition. FLI=% change in fat mass / % change in lean mass + % change in fat mass.
Time Frame: Week 48
Population: All randomized participants who received at least one dose of the study drug and had evaluable data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 55 | 56 | 57 | 55 | 56 | 56 | 55 | 56 | 55
percentage of participants
  >5kg Weight Loss and Fat Loss Index >70 % | 14.55 | 26.79 | 40.35 | 41.82 | 50.00 | 62.50 | 65.45 | 64.29 | 72.73
  >5kg Weight Loss and Fat Loss Index >80 % | 12.73 | 23.21 | 36.84 | 16.36 | 17.86 | 57.14 | 56.36 | 53.57 | 61.82
  >5kg Weight Loss and Fat Loss Index >90 % | 3.64 | 19.64 | 35.09 | 12.73 | 5.36 | 42.86 | 41.82 | 46.43 | 41.82

15. Secondary Outcome: Change From Baseline in Body Fat Mass by Bioelectrical Impedance Analysis (BIA) at Week 48
Description: Body fat was assessed through BIA. LS Mean was determined by ANCOVA model using Baseline + Gender (Male, Female) + Country (Australia, New Zealand, United States of America) + Treatment (Type III sum of squares) as variables. Only participants with non-missing baseline value were included in analysis. Missing values at Week 48 were imputed 100 times based on observed data in the Placebo arm.
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 35 | 31 | 37 | 45 | 51 | 41 | 40 | 43 | 43
kg | -2.78 (1.12) | -5.64 (1.16) | -7.59 (1.01) | -6.95 (0.99) | -10.08 (0.92) | -10.26 (1.03) | -11.72 (1.06) | -11.71 (0.99) | -13.74 (1.00)

16. Secondary Outcome: Change From Baseline in Body Fat Mass by BIA at Week 72
Description: Body fat mass was assessed through BIA.
Time Frame: Baseline, Week 72
Reporting Status: Not Posted, anticipated posting 2026-06

17. Secondary Outcome: Change From Baseline in Body Fat Percentage by BIA at Week 48
Description: Body fat percentage was assessed through BIA. LS Mean was determined by ANCOVA model using Baseline + Gender (Male, Female) + Country (Australia, New Zealand, United States of America) + Treatment (Type III sum of squares) as variables. Only participants with non-missing baseline value were included in analysis. Missing values at Week 48 were imputed 100 times based on observed data in the Placebo arm.
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of body fat
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 55 | 56 | 57 | 55 | 56 | 56 | 55 | 56 | 55
percentage of body fat | -1.69 (0.65) | -3.04 (0.67) | -4.21 (0.61) | -3.42 (0.60) | -4.71 (0.56) | -5.54 (0.62) | -6.77 (0.62) | -6.81 (0.60) | -7.40 (0.59)

18. Secondary Outcome: Change From Baseline in Body Fat Percentage by BIA at Week 72
Description: Body fat percentage was assessed through BIA.
Time Frame: Baseline, Week 72
Reporting Status: Not Posted, anticipated posting 2026-06

19. Secondary Outcome: Change From Baseline in Lean Mass by DXA at Week 48
Description: Lean mass was assessed through DXA. LS Mean was determined by ANCOVA model using Baseline + Gender (Male, Female) + Country (Australia, New Zealand, United States of America) + Treatment (Type III sum of squares) as variables. Only participants with non-missing baseline value were included in analysis. Missing values at Week 48 were imputed 100 times based on observed data in the Placebo arm
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 30 | 30 | 36 | 45 | 47 | 42 | 40 | 42 | 43
kg | -0.5 (0.68) | 0.5 (0.70) | 0.4 (0.65) | -2.6 (0.57) | -3.9 (0.56) | -1.1 (0.63) | -1.2 (0.61) | -0.5 (0.61) | -1.3 (0.58)

20. Secondary Outcome: Change From Baseline in Lean Mass by DXA at Week 72
Description: Lean mass was assessed through DXA.
Time Frame: Baseline, Week 72
Reporting Status: Not Posted, anticipated posting 2026-06

21. Secondary Outcome: Change From Baseline in Lean Body Mass Percentage by DXA at Week 48
Description: Lean body mass percentage was assessed through DXA. LS Mean was determined by ANCOVA model using Baseline + Gender (Male, Female) + Country (Australia, New Zealand, United States of America) + Treatment (Type III sum of squares) as variables. Only participants with non-missing baseline value were included in analysis. Missing values at Week 48 were imputed 100 times based on observed data in the Placebo arm
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of body mass
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 30 | 30 | 36 | 45 | 47 | 42 | 40 | 42 | 43
percentage of body mass | 0.94 (0.69) | 3.38 (0.72) | 5.05 (0.67) | 3.03 (0.65) | 3.81 (0.62) | 5.94 (0.66) | 6.78 (0.67) | 7.13 (0.65) | 8.84 (0.65)

22. Secondary Outcome: Change From Baseline in Lean Body Mass Percentage by DXA at Week 72
Description: DXA was used to assess changes in body composition.
Time Frame: Baseline, Week 72
Reporting Status: Not Posted, anticipated posting 2026-06

23. Secondary Outcome: Change From Baseline in Appendicular Lean Mass by DXA at Week 48
Description: as for outcome 8
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 30 | 30 | 36 | 45 | 47 | 42 | 40 | 42 | 43
kg | -0.3 (0.36) | 0.3 (0.35) | 0.2 (0.34) | -1.2 (0.28) | -2.0 (0.27) | -0.5 (0.30) | -0.6 (0.31) | -0.4 (0.30) | -0.5 (0.28)

24. Secondary Outcome: Change From Baseline in Appendicular Lean Mass by DXA at Week 72
Description: DXA was used to assess changes in body composition.
Time Frame: Baseline, Week 72
Reporting Status: Not Posted, anticipated posting 2026-06

25. Secondary Outcome: Change From Baseline in Lean Mass (kg) by BIA at Week 48
Description: BIA is a widely used method for estimating body composition. LS Mean was determined by ANCOVA model using Baseline + Gender (Male, Female) + Country (Australia, New Zealand, United States of America) + Treatment (Type III sum of squares) as variables. Only participants with non-missing baseline value were included in analysis. Missing values at Week 48 were imputed 100 times based on observed data in the Placebo arm.
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 35 | 31 | 37 | 45 | 51 | 41 | 40 | 43 | 43
kg | -0.71 (0.51) | -0.62 (0.53) | -1.50 (0.51) | -2.97 (0.49) | -3.99 (0.47) | -2.30 (0.50) | -2.50 (0.50) | -2.39 (0.48) | -3.79 (0.50)

26. Secondary Outcome: Change From Baseline in Lean Mass (kg) by BIA at Week 72
Description: BIA is a widely used method for estimating body composition.
Time Frame: Baseline, Week 72
Reporting Status: Not Posted, anticipated posting 2026-06

27. Secondary Outcome: Change From Baseline in Percentage Lean Body Mass by BIA at Week 48
Description: as for outcome 25
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of body mass
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 35 | 31 | 37 | 45 | 51 | 41 | 40 | 43 | 43
percentage of body mass | 2.16 (0.73) | 2.80 (0.80) | 4.17 (0.69) | 3.75 (0.68) | 4.79 (0.64) | 5.42 (0.71) | 6.62 (0.70) | 6.08 (0.67) | 6.95 (0.67)

28. Secondary Outcome: Change From Baseline in Percentage Lean Body Mass by BIA at Week 72
Description: BIA is a widely used method for estimating body composition.
Time Frame: Baseline, Week 72
Reporting Status: Not Posted, anticipated posting 2026-06

29. Secondary Outcome: Percentage of Participants With Body Mass Index (BMI) Categories at Baseline and Week 48
Description: BMI categories:
  i. Healthy weight: 18.5 kilograms (kg)/meter (m)² to 24.9 kg/m² ii. Overweight: 25 kg/m² to 29.9 kg/m² iii. Obesity class 1: 30 kg/m² to 34.9 kg/m² iv. Obesity class II: 35 kg/m² to 39.9 kg/m² v. Obesity class III: ≥ 40 kg/m2
Time Frame: Baseline, Week 48
Population: All randomized participants who received at least one dose of the study drug and had evaluable data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 55 | 56 | 57 | 55 | 56 | 56 | 55 | 56 | 55
percentage of participants
  Healthy weight (Baseline) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Overweight (Baseline) | 1.8 | 5.4 | 1.8 | 14.5 | 5.4 | 3.6 | 9.1 | 1.8 | 5.5
  Obesity class I (Baseline) | 29.1 | 39.3 | 29.8 | 27.3 | 35.7 | 28.6 | 27.3 | 25.0 | 34.5
  Obesity class II (Baseline) | 40 | 30.4 | 38.6 | 27.3 | 32.1 | 30.4 | 29.1 | 50 | 27.3
  Obesity class III (Baseline) | 29.1 | 25 | 29.8 | 30.9 | 26.8 | 37.5 | 34.5 | 23.2 | 32.7
  Healthy weight (Week 48) | 0 | 0 | 2.7 | 17.8 | 3.9 | 2.4 | 10 | 7 | 11.6
  Overweight (Week 48) | 11.4 | 19.4 | 21.6 | 28.9 | 33.3 | 31.7 | 25 | 25.6 | 37.2
  Obesity class I (Week 48) | 37.1 | 32.3 | 43.2 | 17.8 | 51.0 | 31.7 | 37.5 | 53.5 | 27.9
  Obesity class II (Week 48) | 31.4 | 35.5 | 21.6 | 17.8 | 7.8 | 26.8 | 22.5 | 11.6 | 14
  Obesity class III (Week 48) | 20 | 12.9 | 10.8 | 17.8 | 3.9 | 7.3 | 5 | 2.3 | 9.3

30. Secondary Outcome: Percentage of Participants With Baseline Waist-to-Height Ratio (WtHR) Category of <0.5 Having Change From Baseline in Waist-to-Height Ratio (WHtR Ratio) Categories at Week 48
Description: WHtR ratio categories: <0.5; 0.5-0.59; ≥0.6
Time Frame: Baseline up to 48 weeks
Population: All randomized participants who received at least one dose of the study drug and had a baseline WtHR category <0.5 and had evaluable data at week 48.
  As no enrolled participants had a baseline waist-to-height ratio (WtHR) below 0.5, this outcome measure was not analyzed, and no participants were included in the analysis.
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: Percentage of Participants With Baseline WtHR Category of 0.5-0.59 Having Change From Baseline in Waist-to-Height Ratio (WHtR Ratio) Categories at Week 48
Description: WHtR ratio categories: <0.5; 0.5-0.59; ≥0.6
Time Frame: Baseline up to 48 weeks
Population: All randomized participants who received at least one dose of the study drug and had Baseline WtHR Category 0.5-0.59 and had evaluable data at week 48.
  No participants were included in the analysis for the "Bimagrumab 30 mg/kg," "Bimagrumab 10 mg/kg + semaglutide 2.4 mg," and "Bimagrumab 30 mg/kg + semaglutide 1.0 mg" reporting arms, as none of the enrolled individuals in these groups had a baseline WtHR of 0.5-0.59.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 5 | 3 | 0 | 6 | 3 | 2 | 0 | 0 | 4
percentage of participants
  WtHR Category: <0.5 | 0 | 0 |  | 50.0 | 0 | 0 |  |  | 25.0
  WtHR Category: 0.5-0.59 | 60.0 | 100.0 |  | 50.0 | 66.7 | 100.0 |  |  | 75.0
  WtHR Category: ≥0.6 | 40.0 | 0 |  | 0 | 33.3 | 0 |  |  | 0

32. Secondary Outcome: Percentage of Participants With Baseline WtHR Category ≥0.6 Having Change From Baseline in Waist-to-Height Ratio (WHtR Ratio) Categories at Week 48
Description: WHtR ratio categories: <0.5; 0.5-0.59; ≥0.6
Time Frame: Baseline up to 48 weeks
Population: All randomized participants who received at least one dose of the study drug and had Baseline WtHR Category ≥0.6 and had evaluable data at week 48
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 30 | 28 | 37 | 39 | 48 | 39 | 39 | 43 | 39
percentage of participants
  WtHR Category: <0.5 | 0 | 0 | 5.4 | 2.6 | 2.1 | 0 | 7.7 | 2.3 | 15.4
  WtHR Category: 0.5-0.59 | 20.0 | 17.9 | 21.6 | 25.6 | 31.3 | 38.5 | 38.5 | 51.2 | 35.9
  WtHR Category: ≥0.6 | 80.0 | 82.1 | 73.0 | 71.8 | 66.7 | 61.5 | 53.8 | 46.5 | 48.7

33. Secondary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at Week 48
Description: HbA1c is the glycosylated fraction of hemoglobin A. It is measured primarily to identify the average plasma glucose concentration over prolonged periods of time.
Time Frame: Baseline, 48 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 34 | 28 | 33 | 44 | 49 | 40 | 41 | 39 | 43
percentage of HbA1c | -0.0 (0.05) | -0.2 (0.06) | -0.2 (0.05) | -0.3 (0.05) | -0.4 (0.04) | -0.3 (0.05) | -0.5 (0.05) | -0.4 (0.05) | -0.4 (0.05)

34. Secondary Outcome: Change From Baseline in Quality of Life Short Form 36 Version 2 (SF-36v2) Acute Form Physical Functioning Domain Score at Week 24
Description: The SF-36v2 acute form assesses health-related quality of life (HRQoL) on 8 domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. The Physical-Functioning domain assesses limitations due to health "now" and consists of 10-items, each rated on a 3-point Likert scale. Scoring of the domain is norm-based and presented in the form of T-scores, with a mean of 50 and standard deviation of 10; higher scores indicate better levels of function. Range cannot be specified in norm-based scores.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 37 | 38 | 38 | 46 | 46 | 41 | 34 | 39 | 36
t-score | 7.162 (13.720) | 9.211 (11.121) | 14.342 (14.150) | 12.500 (15.230) | 10.435 (14.826) | 12.927 (17.712) | 9.265 (15.132) | 11.667 (18.543) | 17.222 (19.619)

35. Secondary Outcome: Change From Baseline in Quality of Life SF-36v2 Acute Form Total Score Week 24
Description: The SF-36 is a participant-reported outcome measure evaluating participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. The 8 domains are regrouped into (mental component score [MCS] and physical componenet score [PCS] to obtain a total score ranging from 0 to 100, with higher scores indicating better levels of function and/or better health.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 37 | 38 | 38 | 46 | 46 | 41 | 34 | 39 | 36
score on a scale | 6.577 (13.194) | 4.086 (13.219) | 12.193 (13.711) | 13.222 (14.027) | 11.153 (12.357) | 12.124 (16.235) | 7.484 (14.917) | 11.506 (13.528) | 17.060 (13.523)

36. Secondary Outcome: Change From Baseline in Quality of Life SF-36v2 Acute Form Physical Functioning Domain Score Week 48
Description: The SF-36v2 acute form assesses HRQoL on 8 domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. The Physical-Functioning domain assesses limitations due to health "now" and consists of 10 items, each rated on a 3-point Likert scale. Scoring of the domain is norm-based and presented in the form of T-scores, with a mean of 50 and standard deviation of 10; higher scores indicate better levels of function. Range cannot be specified in norm-based scores
Time Frame: Baseline, Week 48
Population: All randomized participants who received at least one dose of the study drug, had a baseline and at least one post- baseline value for this outcome. LS Mean was determined by ANCOVA model using Baseline + Gender(Male, Female) + Country(Australia,New Zealand,United States of America) + Treatment (Type III sum of squares) as variables. Only participants with non-missing baseline value were included in analysis. Missing values at Week 48 imputed 100 times based on observed data in the Placebo arm.
Measure: Least Squares Mean (Standard Error); unit: t-score
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 37 | 38 | 38 | 46 | 46 | 41 | 34 | 39 | 39
t-score | 11.5 (2.14) | 10.8 (2.21) | 12.1 (2.07) | 10.0 (1.91) | 11.6 (1.91) | 14.6 (2.04) | 13.0 (2.06) | 13.0 (2.19) | 16.1 (1.97)

37. Secondary Outcome: Change From Baseline in Quality of Life SF-36v2 Acute Form Total Score at Week 48
Description: The SF-36 is a participant-reported outcome measure evaluating participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. The 8 domains are regrouped into MCS and PCS to obtain a total score ranging from 0 to 100, with higher scores indicating better levels of function and/or better health.
Time Frame: Baseline, Week 48
Population: as for outcome 36
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 37 | 38 | 38 | 46 | 46 | 41 | 34 | 39 | 39
score on a scale | 10.9 (2.26) | 8.5 (2.43) | 11.6 (2.27) | 11.7 (2.01) | 13.5 (1.98) | 14.8 (2.16) | 13.9 (2.25) | 14.4 (2.31) | 16.3 (2.18)

38. Secondary Outcome: Change From Baseline in Quality of Life SF-36v2 Acute Form Physical Functioning Domain Score and Total Score at Week 72
Description: The SF-36v2 acute, 1-week recall version is a 36-item, generic, patient-administered measure designed to assess the following 8 domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. The Physical-Functioning domain assesses limitations due to health "now" while the remaining domains assess functioning "in the past week." Each domain is scored individually and information from these 8 domains are further aggregated into 2 health-component summary scores: Physical-Component Summary and Mental-Component Summary. Items are answered on Likert scales of varying lengths (3-, 5-, or 6- point scales).The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health.
Time Frame: Baseline, Week 72
Reporting Status: Not Posted, anticipated posting 2026-06

39. Secondary Outcome: Change From Baseline in Impact of Weight on Quality of Life-Lite-Clinical Trials Version (IWQOL-Lite-CT) Physical Function Score and Total Score at Week 24
Description: The IWQOL-Lite-CT is a 20-item, obesity-specific PRO instrument developed for use in obesity clinical trials. It assesses 2 primary domains of obesity-related health-related quality of life (HRQoL): physical (7 items) and psychosocial (13 items). Each item is rated on a scale from 0 (worst) to 100 (best), with higher scores indicating better levels of functioning. The IWQOL-Lite-CT provides composite scores for each domain, as well as a total score, all ranging from 0 to 100. Higher scores reflect better levels of functioning and quality of life. This endpoint shows results for 'physical function score' and 'total score.'
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 37 | 38 | 39 | 45 | 47 | 44 | 38 | 42 | 39
score on a scale
  Physical Function Score | 7.973 (15.919) | 13.289 (13.115) | 13.974 (13.726) | 16.667 (14.616) | 17.447 (16.677) | 14.659 (16.474) | 12.105 (22.680) | 18.690 (19.818) | 21.667 (17.113)
  Total score | 8.142 (11.538) | 10.789 (10.363) | 15.513 (11.868) | 17.639 (11.285) | 19.468 (13.055) | 19.468 (13.055) | 14.671 (16.434) | 17.113 (14.463) | 22.917 (14.826)

40. Secondary Outcome: Change From Baseline in IWQOL-Lite-CT Physical Function Score and Total Score at Week 48
Description: as for outcome 39
Time Frame: Baseline, Week 48
Population: as for outcome 36
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
Number analyzed (Participants) | 34 | 29 | 35 | 43 | 45 | 40 | 37 | 36 | 39
score on a scale
  Physical Function Score | 13.3 (2.65) | 15.6 (2.71) | 16.1 (2.62) | 15.3 (2.41) | 19.5 (2.33) | 18.7 (2.57) | 19.3 (2.53) | 21.6 (2.58) | 20.2 (2.39)
  Total Score | 14.1 (2.42) | 14.7 (2.36) | 16.6 (2.40) | 17.5 (2.19) | 21.6 (2.17) | 22.4 (2.26) | 19.2 (2.33) | 21.2 (2.38) | 23.8 (2.22)

41. Secondary Outcome: Change From Baseline in IWQOL-Lite-CT Physical Function Score and Total Score at Week 72
Description: as for outcome 39
Time Frame: Baseline, Week 72
Reporting Status: Not Posted, anticipated posting 2026-06

ADVERSE EVENTS:
Time Frame: Baseline up to Week 48
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
  Safety data from the Open Label Extension Treatment Period (Weeks 49 to 72) and Post-Treatment Follow-Up Period (Weeks 73 to 104) will be reported during the final results posting, i.e., no later than June, 2026.
Arm/Group | Placebo | Bimagrumab 10 mg/kg | Bimagrumab 30 mg/kg | Placebo + Semaglutide 1.0 mg | Placebo + Semaglutide 2.4 mg | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/56 | 0/57 | 0/55 | 0/56 | 0/56 | 0/55 | 0/56 | 0/55
Serious Adverse Events (participants affected / at risk) | 2/55 | 7/56 | 5/57 | 1/55 | 6/56 | 4/56 | 5/55 | 2/56 | 3/55
Other Adverse Events (participants affected / at risk) | 41/55 | 52/56 | 53/57 | 52/55 | 51/56 | 52/56 | 54/55 | 54/56 | 54/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=55) | Bimagrumab 10 mg/kg (N=56) | Bimagrumab 30 mg/kg (N=57) | Placebo + Semaglutide 1.0 mg (N=55) | Placebo + Semaglutide 2.4 mg (N=56) | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg (N=56) | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg (N=55) | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg (N=56) | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg (N=55)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder enlargement (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perineal cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/31 (0) | 1/32 (1) | 0/33 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=55) | Bimagrumab 10 mg/kg (N=56) | Bimagrumab 30 mg/kg (N=57) | Placebo + Semaglutide 1.0 mg (N=55) | Placebo + Semaglutide 2.4 mg (N=56) | Bimagrumab 10 mg/kg + Semaglutide 1.0 mg (N=56) | Bimagrumab 10 mg/kg + Semaglutide 2.4 mg (N=55) | Bimagrumab 30 mg/kg + Semaglutide 1.0 mg (N=56) | Bimagrumab 30 mg/kg + Semaglutide 2.4 mg (N=55)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oestrogen deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extraocular muscle disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital dermatitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Posterior capsule opacification (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 9 (9) | 1 (1) | 6 (6) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 5 (5) | 8 (8) | 7 (7) | 5 (5) | 8 (8)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 8 (8) | 2 (2) | 3 (3)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 11 (11) | 16 (16) | 8 (8) | 15 (15) | 15 (15) | 9 (9)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 23 (23) | 28 (28) | 19 (19) | 20 (20) | 24 (24) | 29 (29) | 24 (24) | 26 (26)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 6 (6) | 4 (4) | 5 (5) | 3 (3) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 5 (5) | 1 (1) | 2 (2)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 5 (5) | 3 (3) | 3 (3) | 8 (8) | 5 (5) | 6 (6)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal metaplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 14 (14) | 7 (7) | 25 (25) | 26 (26) | 23 (23) | 34 (34) | 21 (21) | 27 (27)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tongue spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (3) | 5 (5) | 9 (9) | 6 (6) | 10 (10) | 6 (6) | 7 (7)
Administration site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Exercise tolerance decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 3 (3) | 4 (4) | 12 (12) | 14 (14) | 5 (5) | 12 (12) | 7 (7) | 12 (12)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 5 (5) | 3 (3) | 2 (2) | 4 (4) | 1 (1)
Infusion site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Oedema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immunisation reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Acne pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Covid-19 (Infections and infestations) | 8 (8) | 13 (13) | 10 (10) | 12 (12) | 16 (16) | 10 (10) | 3 (3) | 3 (3) | 9 (9)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Ear infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gonorrhoea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 6 (6) | 2 (2) | 4 (4) | 5 (5) | 4 (4) | 2 (2) | 4 (4) | 2 (2)
Omphalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post viral fatigue syndrome (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-acute covid-19 syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pustule (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 12 (12) | 11 (11) | 11 (11) | 12 (12) | 8 (8) | 7 (7) | 11 (11) | 11 (11)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 5 (5) | 5 (5) | 5 (5) | 5 (5)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0/31 (0) | 0/32 (0) | 0/33 (0) | 2/32 (2) | 0/32 (0) | 0/32 (0) | 1/32 (1) | 0/32 (0) | 0/32 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/31 (0) | 0/32 (0) | 0/33 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 1/32 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burn oral cavity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body in skin or subcutaneous tissue (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 5 (5) | 3 (3)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 6 (6) | 8 (8) | 7 (7) | 3 (3) | 1 (1) | 6 (6) | 9 (9) | 8 (8) | 7 (7)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood folate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone density decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram t wave inversion (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Human metapneumovirus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 2 (2) | 3 (3) | 5 (5) | 6 (6) | 1 (1) | 5 (5) | 3 (3) | 2 (2)
Lipids increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nitrite urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic enzymes increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Red blood cell sedimentation rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Red blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urine bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vitamin b12 decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 4 (4) | 6 (6) | 7 (7) | 10 (10) | 6 (6) | 8 (8) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 6 (6) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 6 (6) | 4 (4) | 5 (5) | 3 (3) | 2 (2)
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exostosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 26 (26) | 42 (42) | 7 (7) | 5 (5) | 32 (32) | 35 (35) | 34 (34) | 35 (35)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 3 (3) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 7 (7) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 3 (3) | 1 (1) | 2 (2) | 5 (5) | 2 (2) | 4 (4) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allodynia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4) | 2 (2) | 2 (2) | 7 (7) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 7 (7)
Headache (Nervous system disorders) | 6 (6) | 11 (11) | 6 (6) | 10 (10) | 10 (10) | 9 (9) | 12 (12) | 12 (12) | 9 (9)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hyporeflexia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Migraine with aura (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Radicular pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thoracic radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue biting (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysphoria (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Grief reaction (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Negative thoughts (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parasomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Albuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sterile pyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0/31 (0) | 0/32 (0) | 0/33 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 1/32 (1) | 0/32 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0/31 (0) | 0/32 (0) | 0/33 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 1/32 (1) | 0/32 (0) | 0/32 (0)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 1/31 (1) | 0/32 (0) | 0/33 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 1/32 (1) | 0/32 (0)
Endometriosis (Reproductive system and breast disorders) | 0/31 (0) | 0/32 (0) | 0/33 (0) | 0/32 (0) | 1/32 (1) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/23 (0) | 0/24 (0) | 1/24 (1) | 0/23 (0) | 0/24 (0) | 0/23 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/23 (0) | 0/24 (0) | 0/24 (0) | 0/23 (0) | 1/24 (1) | 0/23 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0/31 (0) | 0/32 (0) | 1/33 (1) | 1/32 (1) | 2/32 (2) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0/31 (0) | 0/32 (0) | 0/33 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 2/32 (2) | 0/32 (0) | 0/32 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0/31 (0) | 0/32 (0) | 0/33 (0) | 0/32 (0) | 1/32 (1) | 0/32 (0) | 0/32 (0) | 1/32 (1) | 0/32 (0)
Menstrual disorder (Reproductive system and breast disorders) | 1/31 (1) | 0/32 (0) | 0/33 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0)
Menstruation delayed (Reproductive system and breast disorders) | 0/31 (0) | 0/32 (0) | 0/33 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 1/32 (1) | 0/32 (0) | 0/32 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0/31 (0) | 0/32 (0) | 0/33 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 2/32 (2) | 0/32 (0) | 0/32 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0/31 (0) | 1/32 (1) | 0/33 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0)
Ovarian disorder (Reproductive system and breast disorders) | 0/31 (0) | 0/32 (0) | 0/33 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 1/32 (1) | 0/32 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0/31 (0) | 1/32 (1) | 1/33 (1) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0)
Testicular pain (Reproductive system and breast disorders) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/23 (0) | 0/24 (0) | 0/24 (0) | 0/23 (0) | 0/24 (0) | 0/23 (0)
Uterine polyp (Reproductive system and breast disorders) | 0/31 (0) | 0/32 (0) | 1/33 (1) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0/31 (0) | 0/32 (0) | 0/33 (0) | 1/32 (1) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0/31 (0) | 0/32 (0) | 1/33 (1) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/31 (0) | 0/32 (0) | 0/33 (0) | 1/32 (1) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinonasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 19 (19) | 25 (25) | 6 (6) | 5 (5) | 24 (24) | 25 (25) | 31 (31) | 29 (29)
Acne cystic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Androgenetic alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chloasma (Skin and subcutaneous tissue disorders) | 0/31 (0) | 0/32 (0) | 0/33 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 1/32 (1) | 0/32 (0) | 0/32 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 0/31 (0) | 0/32 (0) | 0/33 (0) | 0/32 (0) | 1/32 (1) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Keloid scar (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 3 (3)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (7) | 1 (1) | 4 (4) | 2 (2) | 8 (8) | 5 (5) | 5 (5) | 5 (5)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abstains from alcohol (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcohol use (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menopause (Social circumstances) | 0/31 (0) | 1/32 (1) | 0/33 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0) | 0/32 (0)
Lipoma excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angiopathy (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein ruptured (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT05616013/Prot_002.pdf
  • Statistical Analysis Plan (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT05616013/SAP_003.pdf